CLINICAL TRIAL: NCT00959296
Title: Implantable Systems Performance Registry
Acronym: ISPR
Status: Completed | Type: Observational
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Other Study IDs: NSP0010-10000
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Spinal Cord Stimulation; Deep Brain Stimulation; Drug Infusion (Implantable Pumps); Sacral Neuromodulation
Keywords: Registry; Pain; Chronic Pain; Back Pain; Intractable Spasticity; Parkinson's Disease; Essential Tremor; Dystonia; Implantable Pumps; Incontinence
MeSH Terms: conditions — Pain; Chronic Pain; Back Pain; Parkinson Disease; Essential Tremor; Dystonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with a device implant: Patients implanted and consented at a study center with a market-released Medtronic implantable drug pump, spinal cord stimulator, deep brain stimulator, or sacral nerve stimulator.
  Interventions: Device: Various

INTERVENTIONS:
Device: Various — Patients implanted and consented at a study center with a market-released Medtronic implantable drug pump, spinal cord stimulator, deep brain stimulator, or sacral nerve stimulator.

SUMMARY:
The Implantable Systems Performance Registry (ISPR) was developed to evaluate the long-term reliability and performance of market-released Medtronic Neuromodulation infusion and stimulation products.

Completion Notice: The ISPR was created by Medtronic to monitor the performance of commercially available products. This registry was initially designed to track performance of Medtronic's implantable infusion and spinal cord stimulation systems beginning in August 2003 and June 2004, respectively. Medtronic DBS Systems were added to the ISPR in June 2009, and Sacral Neuromodulation Systems in April 2010. Medtronic retired the ISPR in April 2016 and merged the data collected from this registry into the Product Surveillance Registry (PSR). Please refer to that record, Clinical Trials identifier: NCT01524276, for further information.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for an implant or replacement with a market-released Medtronic implantable drug pump, spinal cord stimulator, deep brain stimulator, or sacral nerve stimulator

Exclusion Criteria:

* Patient who is or will be inaccessible for follow-up at an ISPR study site
* Patient is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound the results of this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 10981 (Actual)
Dates: Start 2003-08; Primary Completion 2016-09-27 (Actual); Study Completion 2016-09-27 (Actual)

PRIMARY OUTCOMES:
Product Performance | Annually
  To quantify and compare the rates of device-related events for market-released Medtronic Neuromodulation infusion and stimulation devices

CONTACTS AND LOCATIONS:
Overall Officials: ISPR Team, Study Chair — Medtronic
Locations (50):
- United States (43):
  - Huntsville, Alabama
  - Scottsdale, Arizona
  - Aliso Viejo, California
  - Los Angeles, California
  - Napa, California
  - Palm Springs, California
  - Pasadena, California
  - San Diego, California
  - Upland, California
  - Washington D.C., District of Columbia
  - Site recruiting for sacral nerve stimulation, Bradenton, Florida
  - Merritt Island, Florida
  - Ocala, Florida
  - Atlanta, Georgia
  - Gainesville, Georgia
  - Bloomington, Illinois
  - Chicago, Illinois
  - Evansville, Indiana
  - Muncie, Indiana
  - South Bend, Indiana
  - Iowa City, Iowa
  - West Des Moines, Iowa
  - Annapolis, Maryland
  - Silver Spring, Maryland
  - Westminster, Maryland
  - Minneapolis, Minnesota
  - Saint Paul, Minnesota
  - St Louis, Missouri
  - Buffalo, New York
  - Great Neck, New York
  - New York, New York
  - Poughkeepsie, New York
  - Winston-Salem, North Carolina
  - Site is recruiting for Deep Brain Stimulation, Cincinnati, Ohio
  - West Chester, Ohio
  - York, Pennsylvania
  - Nashville, Tennessee
  - Houston, Texas
  - Tyler, Texas
  - Salt Lake City, Utah
  - Roanoke, Virginia
  - Bremerton, Washington
  - Seattle, Washington
- Vienna, Austria
- Montpellier, France
- Germany (2):
  - Cologne
  - Hanover
- Pavia, Italy
- Barcelona, Spain
- Oxford, United Kingdom